CLINICAL TRIAL: NCT03750188
Title: The Safety and Efficacy of ProHance® at the Dose of 0.10 mmol/kg in Magnetic Resonance Imaging of the Central Nervous System in Pediatric Patients Who Are Younger Than 2 Years of Age
Brief Title: Evaluation of Safety and Efficacy of ProHance in Pediatric Patients <2yrs
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PH-108
Record Dates: First submitted 2018-11-07; First posted 2018-11-21 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2018-11

CONDITIONS: Central Nervous System Diseases; Central Nervous System Neoplasms
Keywords: CNS; MRI; ProHance; Gadoteridol
MeSH Terms: conditions — Central Nervous System Diseases; Central Nervous System Neoplasms | interventions — gadoteridol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: ProHance — 0.1 mmol/kg ProHance intravenous injection
  Other Names: Gadoteridol

SUMMARY:
Safety and Efficacy Study in pediatric subjects <2 years of age who have undergone Brain or Spine MRI pre and post 0.1 mmol/kg ProHance administration. Imaging conditions will represent those in routine clinical practice. Retrospective enrolment with a prospective blinded read.

DETAILED DESCRIPTION:
The purpose of this study is to retrospectively enroll children younger than 2 years of age who have undergone brain or spine MRI with 0.1 mmol/kg PROHANCE and to gather safety data as well as to collect MR images for a prospective blinded read to evaluate the efficacy of PROHANCE in terms of visualization and enhancing properties.

The study will be conducted in 4-8 sites in the United States and Europe. It is estimated that 120 patients will be enrolled to provide 108 evaluable patients.

Three radiologists unaffiliated with enrolling centers (blinded readers), blinded to the patient's identity and clinical profile will independently evaluate the MRI images. The efficacy analysis will be primarily based on the blinded reader evaluations.

Imaging conditions will represent those in routine clinical practice, inclusive of pre and post-contrast images.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female and was younger than 2 years of age at the time of the MRI with PROHANCE injection at the dose of 0.1 mmol/kg (±25% in volume administered).
* Has demographic information, reason for the ProHance-enhanced MR examination, relevant medical history, final diagnosis, and safety data available.
* Has documented known or highly suspected enhancing disease of CNS (brain/spine) and previously underwent a cranial or spinal MR examination requiring an injection of PROHANCE contrast agent.
* Has both predose and postdose T1 SE/FSE and/or GRE and T2 SE/FSE, and FLAIR MR images (when available) for submission to Bracco or designee to be evaluated in a fully blinded read.
* Has complete information on the imaging protocol used for the ProHance-enhanced MR exam including type of exam (brain or spine), MR scanner and field strength (1.0, 1.5 or 3.0 Tesla)
* Has a documented dose of PROHANCE administered for their MRI exam and/or the volume (mL) and weight of the patient available to be used to calculate the exact dose of PROHANCE that was administered.

Exclusion Criteria:

• Exclude a patient from this study if the patient does not fulfill all of the inclusion criteria.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will include patients younger than 2 years of age who have previously undergone MRI of the CNS (brain or spine) with PROHANCE at the dose of 0.1 mmol/kg as part of their clinical work-up.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Border delineation of lesions | Immediately post dose - Day 1
  Blinded reader will assess the border delineation of lesion based on a 5 point scale, none (0) - Excellent (4)
Visualization of internal morphology of lesions | Immediately post dose - Day 1
  Blinded reader will assess the visualization of internal morphology of the lesion(s) based on a 5 point scale, none (0) - Excellent (4)
Contrast enhancement of lesions | Immediately post dose- Day 1
  Blinded reader will assess the contrast enhancement of the lesion(s) based on a 5 point scale, none (0) - Excellent (4)
Number and percentage of subjects with ProHance Related Adverse Events | up to 2 hours post-dose
  In terms of frequency, type and severity of adverse events Data collected, will consist of Screening Serum Creatinine value (mg/dL), If available, Vital signs (systolic blood pressure, diastolic blood pressure, heart rate, respiration rate) and ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No